CLINICAL TRIAL: NCT06869018
Title: A Randomized, Investigator- and Participant-blinded, Multiple-ascending Dose, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3549492 in Japanese Participants With Type 2 Diabetes Mellitus and Healthy Japanese Participants
Brief Title: A Study of LY3549492 in Japanese Participants With Type 2 Diabetes Mellitus (T2D) and Healthy Japanese Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27338; J3H-JE-GZNG (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-10; First posted 2025-03-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Type 2 Diabetes Mellitus (T2D)
Keywords: Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3549492 Part A (Experimental): LY3549492 administered orally
  Interventions: Drug: LY3549492
- LY3549492 Part B (Experimental): LY3549492 administered orally
  Interventions: Drug: LY3549492
- Placebo Part A (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- Placebo Part B (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3549492 — Administered orally
  Arms: LY3549492 Part A; LY3549492 Part B
Drug: Placebo — Administered orally
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of this study is to evaluate how well LY3549492 is tolerated and what side effects may occur in Japanese participants with Type 2 Diabetes Mellitus (T2D) and healthy Japanese participants. The study drug will be administered orally. Blood tests will be performed to check how much LY3549492 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 19 weeks for both Part A (Cohorts 1-3) for multiple-ascending doses (MAD), and Part B (Cohorts 4-5) multiple-ascending doses (MAD), for a total of approximately 25 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Participants with T2DM for at least 6 months
* With an HbA1c value:

  * equal to or greater than 7.0% and equal to or less than 10.0% at screening for participants treated with diet and exercise alone, OR
  * equal to or greater than 6.5% and equal to or less than 9.0% for participants prior to washout of antidiabetic medications
* Have had a stable weight for the 3 months prior to screening. Stable weight is defined as less than 5% body weight change

Part B:

* Have safety laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator. Laboratory tests may be repeated if there is a documented technical error, or once at the discretion of the investigator for any out-of-range results

Exclusion Criteria:

* Have a known clinically significant gastric emptying abnormality
* Have a 12-lead electrocardiogram (ECG) abnormality
* Have an abnormal blood pressure or pulse rate
* Have a significant history within the past 6 months or current evidence of comorbidities capable of altering the absorption, metabolism, or elimination of drug. Or constituting a risk when taking the study drug
* Have a history of chronic medical conditions involving the heart, liver, or kidneys

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Day 1 Through Day 127
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3549492 | Day 1 Through Day 127
  PK: AUC of LY3549492
PK: Maximum Concentration (Cmax) of LY3549492 | Day 1 Through Day 127
  PK: Cmax of LY3549492
Pharmacodynamic (PD): Part A: Change from Baseline in Hemoglobin A1c (HbA1c) | Day 1 Through Day 127
  PD: Change from Baseline in Hemoglobin A1c (HbA1c)
PD: Change from Baseline in Body Weight | Day 1 Through Day 127
  PD: Change from Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - Hakata Clinic, Fukuoka
  - P-One Clinic, Hachiōji
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka
  - Clinical Research Hospital Tokyo, Shinjuku-ku

IPD SHARING:
Plan to Share IPD: No